CLINICAL TRIAL: NCT05882734
Title: An Open Label, Multicenter, Phase 1b/2a Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of the ATR Inhibitor M1774 in Combination With Cemiplimab in Participants With Non-Squamous Non-Small Cell Lung Cancer That Has Progressed on Prior Anti-PD-(L)1 and Platinum-based Therapies (DDRiver NSCLC 322)
Brief Title: Tuvusertib (M1774) in Combination With Cemiplimab in Participants With Non-Squamous NSCLC (DDRiver NSCLC 322)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201924_0022; 2022-502010-85-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Ataxia telangiectasia mutated and Rad3-related protein kinase (ATR) inhibitor; Tuvusertib (M1774); Non squamous Non small cell lung cancer; Cemiplimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Hereditary Sensory and Autonomic Neuropathies | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dosing Regimen 1 (Phase 1b): M1774 + Cemiplimab (Experimental)
  Interventions: Drug: M1774; Drug: Cemiplimab
- Dosing Regimen 2 (Phase 1b): M1774 + Cemiplimab (Experimental)
  Interventions: Drug: M1774; Drug: Cemiplimab
- Stratum A (Phase 2a): Either Dosing Regimen 1 or 2 as finalized in Phase 1b (Experimental)
  Interventions: Drug: M1774; Drug: Cemiplimab
- Stratum B (Phase 2a): Either Dosing Regimen 1 or 2 as finalized in Phase 1b (Experimental)
  Interventions: Drug: M1774; Drug: Cemiplimab
- Stratum C (Phase 2a): Either Dosing Regimen 1 or 2 as finalized in Phase 1b (Experimental)
  Interventions: Drug: M1774; Drug: Cemiplimab

INTERVENTIONS:
Drug: M1774 — In Phase 1b, M1774 will be administered as dosing regimen 1 or dosing regimen 2 until disease progression, death discontinuation criteria or any other reason. The selected dosing regimen of M1774 will be administered in all arms of Phase 2a.
  Other Names: Tuvusertib
Drug: Cemiplimab — Cemiplimab will be administered as an intravenous infusion every 3 weeks in all arms of Phase 1b and Phase 2a until disease progression, death discontinuation criteria or any other reason.

SUMMARY:
This is an Open-label, multicenter clinical study conducted in two Phases to establish the efficacy, safety, tolerability, and pharmacokinetics of the ataxia telangiectasia mutated and Rad3-related protein kinase (ATR) inhibitor Tuvusertib in Combination with Cemiplimab in Participants with Non-Squamous Non-Small Cell Lung Cancer (nsqNSCLC) that has Progressed on Prior Anti-PD-(L)1 and Platinum-based Therapies..

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with nsqNSCLC histologically or cytologically confirmed
* Participants with Radiologically confirmed/documented disease progression during or after the following systemic therapies (all required):

  * At most, 1 line of anti-PD-(L)1 therapy for locally advanced or metastatic disease. Rechallenge with the same anti-PD-(L)1 for disease considered sensitive to anti-PD-(L)1 therapy (e.g. after a treatment break) is considered 1 line
  * Platinum-based therapy for locally advanced or metastatic disease, given in combination or sequentially with anti-PD-(L)1 therapy. Participants who received adjuvant platinum-based therapy meet this criterion if disease progression occurred within 6 months from the last dose that the participant received that therapy. No additional cytotoxic therapies after progression on platinum-based therapy are allowed
  * Prior best overall response of stable disease or better with anti-PD-(L)1 therapy
  * Disease progression must have occurred while the participant has been receiving anti-PD-(L)1 therapy or within 16 weeks of the last dose of anti-PD-(L)1 therapy
* Participants with Measurable disease per RECIST v1.1
* Participants with Eastern Cooperative Oncology Group (ECOG) PS 0 or 1
* Adequate hematological, hepatic, and renal function as defined in the protocol.
* Phase 2a part only: central liquid biopsy analysis of tumor molecular alterations with an assay with appropriate regulatory status
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants with tumors harboring actionable epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) genomic aberrations. Participants with tumors with other actionable aberrations are eligible and allowed to have received up to 1 line of available targeted therapy
* Participants with history of additional malignancy within 3 years before the date of enrollment. Exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the Investigator, with concurrence of the Sponsor's Medical Monitor, is considered cured with minimal risk of recurrence within 3 years
* Participants with known brain metastases, unless clinically stable
* Participant with history of (noninfectious) pneumonitis that required systemic corticosteroids or current pneumonitis/interstitial lung disease
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1b/Phase 2a: Confirmed Overall response (OR) According to Response Evaluation Criteria in Solid Tumor (RECIST) 1.1 As assessed by Investigator | Time from randomization to final assessment or until progression disease, death, discontinuation criteria approximately up to 3 years and 2 months
Phase 1b: Number of Participants With Adverse Events (AEs) and Treatment-related AEs | Time from randomization to final assessment at end of safety follow-up visit approximately up to 3 years and 2 months

SECONDARY OUTCOMES:
Phase 1b/Phase 2a: Duration of Response (DoR) According to RECIST 1.1 as Assessed by the Investigator | Time from randomization to final assessment or until progression disease, death, discontinuation criteria approximately up to 3 years and 2 months
Phase 1b/Phase 2a: Progression Free Survival (PFS) According to RECIST 1.1 as Assessed by the Investigator | Time from randomization to final assessment or until progression disease, death, discontinuation criteria approximately up to 3 years and 2 months
Phase 1b/Phase 2a: Overall survival (OS) | Time from randomization to final assessment or until progression disease, death, discontinuation criteria approximately up to 3 years and 2 months
Phase 2a: Number of Participants With AEs and Treatment-related AEs | Time from randomization to final assessment at end of safety follow-up visit (approximately up to 3 years and 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (54):
- United States (6):
  - UCLA Hematology and Oncology - Santa Monica, Santa Monica, California
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Cancer Specialists - Biomedical Research, Knoxville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Research & Clinical Development, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Belgium (6):
  - Institut Jules Bordet - Department of Institut Jules Bordet', Anderlecht
  - UZA - Oncology, Edegem
  - Jessa Ziekenhuis Hospital, Hasselt
  - Universitair Ziekenhuis Brussel - UZB, Jette
  - UZ Leuven, Leuven
  - CHU de Liège - PARENT, Liège
- France (7):
  - CHU Angers - Hôpital Larrey - Service de Pneumologie, Angers
  - Centre Hospitalier Intercommunal de Créteil - Service de Pneumologie, Créteil
  - CHU Limoges - Hôpital Dupuytren - Unite d'Oncologie Thoracique et Cutanée, Limoges
  - Hôpital de la Timone - CPCEM CIC - Bat F 1er étage, Marseille
  - Hopital Arnaud de Villeneuve - Service de Pneumologie-Addictologie, Montpellier
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Unité d'Explorations Fonctionnelles Respiratoires, Pessac
  - ICO - Site René Gauducheau - Service d'Oncologie medicale, Saint-Herblain
- Germany (3):
  - Universitaetsklinikum Giessen und Marburg GmbH - Medizinische Klinik und Poliklinik III, Giessen
  - Universitaetsklinikum Leipzig AoeR - Med. Klinik u. Poliklinik I - Abt. Pneumologie, Leipzig
  - Sana Klinikum Offenbach GmbH - Medizinische Klinik IV, Offenbach
- Italy (7):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS - U.O. Oncologia Medica, Bologna
  - IEO Istituto Europeo di Oncologia - Divisione Oncologia Medica, Milan
  - Ospedale San Raffaele - U.O. di Oncologia Medica, Milan
  - Istituto Nazionale Tumori Fondazione G. Pascale - Medical Oncology Thoraco-Pulmonary Department, Napoli
  - Istituto Nazionale Tumori Regina Elena IRCCS - S.C. Oncologia Medica B, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Rome
  - Istituto Clinico Humanitas - U.O. di Oncologia Medica ed Ematologia, Rozzano
- Japan (8):
  - National Cancer Center Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata-shi
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of JFCR, Kōtoku
  - Kurume University Hospital, Kurume-shi
  - Aichi Cancer Center Hospital, Nagoya
  - Kindai University Hospital, Osakasayama-shi
  - Kanagawa Cancer Center, Yokohama
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System - Division of Infectious Diseases, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (13):
  - Hospital Clinic de Barcelona - Servicio de Oncologia, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - Hospital Universitario Reina Sofia - Dept of Oncology, Córdoba
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital Universitario 12 de Octubre - Servicio de Oncologia, Madrid
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz - Oncology Department, Madrid
  - Hospital Universitario Ramon y Cajal - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga - Oncology Dept, Málaga
  - Hospital Universitario Nuestra Señora de Valme - Servicio de Oncologia, Seville
  - Hospital Universitario Virgen del Rocio - Oncology Service, Seville
  - Hospital Universitario Virgen Macarena - Oncology Service, Seville
  - Hospital Universitari i Politecnic La Fe - Oncology Department, Valencia

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201924_0022
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html